CLINICAL TRIAL: NCT04365452
Title: Medela INVIA Motion NPWT System for Prophylactic Use on Surgical Incision After Cesarean Delivery
Brief Title: The Invia Motion at Cesarean Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Medela AG (Industry)
Responsible Party: Principal Investigator, David Haas, Professor of Obstetrics and Gynecology, Indiana University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HC#1902
Record Dates: First submitted 2020-03-05; First posted 2020-04-28 (Actual); Results first posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Negative Pressure Wound Therapy; Cesarean Section; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Medela Invia pump
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Invia Motion Arm (Experimental)
  Interventions: Device: Invia Motion

INTERVENTIONS:
Device: Invia Motion — Invia Motion NPWT system at cesarean delivery

SUMMARY:
To assess patient centered outcomes of the Medela INVIA Motion prophylactic NPWT system at cesarean delivery.

DETAILED DESCRIPTION:
This study will be a two center case series of women undergoing caesarean delivery conducted at two medical centers in Indianapolis, Indiana.

All patients meeting inclusion criteria will be included. All enrolled patients will receive the Medela INVIA Motion prophylactic NPWT device.

Visit A: Interventional Procedure All enrolled patients will receive the Medela INVIA Motion device placed by the patient's surgeon after the skin is closed with subcuticular suture or staples. Research staff and clinicians (labor & delivery and postpartum nurses, OR technicians, physicians, etc.) involved in the study will receive formal training on how to place and remove the prophylactic NPWT device.

Visit B: Post Procedure until Discharge Patients will be monitored daily while in the hospital by clinical staff and/or research staff for complications.

The negative pressure wound therapy dressing will be removed on the day of discharge. If the patient remains hospitalized for more than 7 days, the dressing will be removed on postoperative day 7.

Replacement of any dressing that is saturated. If a patient develops infection with the NPWT device in place the device will be removed and the patient given standard SSI therapy as outlined below.

Patients will be educated about the signs and symptoms of infection and other study outcomes and encouraged to call their provider if these should arise.

Research staff document inpatient course regarding SSI. Management of surgical site infections will follow the Practice Guidelines of the Infectious Diseases Society of America.

Visit C: Postpartum Follow Up

We will use active surveillance by research staff to ascertain surgical site infections:

Research staff will follow-up with the research participant at time of discharge or within 48 hours post discharge (postpartum day 1-9) to assess for adverse events, assess the participant's pain, obtain their satisfaction with their dressing and aesthetic appearance of the incision.

Research staff will call subjects on approximately postoperative day 30 (±2 days). They will ask the patient standardized questions regarding wound complications, patient satisfaction, pain and aesthetic appearance. If the patient reports a hospital, clinic, or ER visit not associated with the study centers, the staff will obtain the name of the medical facility and request the records.

The EQ-5D-3L quality of life questionnaire will be administered at the 30-day call.

Medical records from postpartum clinic visits as well as records of unscheduled visits (to any hospital clinic or ER) will be sought to ascertain study outcomes.

At the time of the subject's standard of care postpartum appointment about 4-6 weeks after inpatient hospital discharge research staff will collect information on outcomes, pain and patient satisfaction. If the patient does not attend the clinical postpartum visit, the study staff will contact the subject by phone to collect the data.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled/non-labor or unscheduled/labor cesarean delivery
2. Gestational age greater than or equal to 23 weeks

Exclusion Criteria:

1. Unwilling or unable to provide consent
2. Non-availability for postoperative follow-up
3. Contraindication to NPWT

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Methodius Tuuli, MD, MPH, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patient undergoing cesarean delivery who consented were included
Period: Overall Study
Arm/Group | Invia Motion Arm
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25 [22 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores: Discharge Time Frame
Description: Pain scores (pain score on scale of 0 - 10); 0 represents no pain, 10 represents highest pain
Time Frame: At post-operative day 3 (+/- 1 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
score on a scale | 2.5 [1 to 5]

2. Primary Outcome: Pain Scores: Scores Postpartum Day 30
Description: Pain scores (pain score on scale of 0 - 10); 0 represents no pain, 10 represents highest pain
Time Frame: At postoperative day 30 (+/- 2 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
score on a scale | 0 [0 to 1]

3. Primary Outcome: Patient Satisfaction: Scores Discharge Time Frame
Description: Patient satisfaction scores (satisfaction score on scale of 0 - 10); 0 represents no satisfaction, 10 represents highest satisfaction
Time Frame: At postoperative day 3 (+/- 1 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
score on a scale | 10 [8.5 to 10]

4. Primary Outcome: Patient Satisfaction: Scores Postpartum Day 30
Description: as for outcome 3
Time Frame: At postoperative day 30 (+/- 2 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
score on a scale | 10 [10 to 10]

5. Primary Outcome: Patient Satisfaction With Aesthetic Appearance: Scale
Description: Patient satisfaction with aesthetic appearance (satisfaction score on scale of 0 - 10); 0 represents no satisfaction, 10 represents highest satisfaction
Time Frame: At postoperative day 30 (+/- 2 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
score on a scale | 10 [10 to 10]

6. Secondary Outcome: Wound Infection; Proportion of Incidence
Description: Composite wound complication; wound infection as diagnosed by treating clinician
Time Frame: 4-6 Weeks Postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
Participants | 0

7. Secondary Outcome: Wound Separation; Proportion of Incidence
Description: Composite wound complication; wound separation as diagnosed by treating clinician
Time Frame: 4-6 Weeks Postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
Participants | 0

8. Secondary Outcome: Seroma; Proportion of Incidence
Description: Composite wound complication; seroma as diagnosed by treating clinician
Time Frame: 4-6 Weeks Postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
Participants | 0

9. Secondary Outcome: Antibiotics Prescribed for Presumed SSI; Proportion of Incidence
Description: Composite wound complication; antibiotics prescribed by treating clinician for wound-related infection
Time Frame: 4-6 Weeks Postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
Participants | 0

10. Secondary Outcome: Skin Blistering; Safety Outcomes
Description: Safety outcome; proportion of incidence of skin blistering around surgical wound
Time Frame: 4-6 Weeks Postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
Participants | 0

11. Secondary Outcome: Allergic Reaction; Safety Outcomes
Description: Safety outcome; proportion of allergic reaction to wound dressing
Time Frame: 4-6 Weeks Postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
Participants | 0

12. Secondary Outcome: Wound Bleeding; Safety Outcomes
Description: Safety outcome; proportion of wound bleeding
Time Frame: 4-6 Weeks Postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Invia Motion Arm
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: 4 - 6 weeks
Arm/Group | Invia Motion Arm
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT04365452/Prot_SAP_001.pdf